CLINICAL TRIAL: NCT04380233
Title: A Multi-center, Randomized, Double-Blind, Placebo-Controlled Parallel Group Clinical Research of Zhizhu Kuanzhong Capsule in Treating Patients With Functional Dyspepsia-Postprandial Distress Syndrome
Brief Title: Zhizhu Kuanzhong Capsule for Patients With Functional Dyspepsia-Postprandial Distress Syndrome
Acronym: ZZKZ-FD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhong Lidan, Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HKBU-FD
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Drugs, Investigational; Drug Evaluation

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Parallel Group Clinical Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The eligible subjects will be randomly assigned, with equal access to either the Chinese medicine treatment investigational drug group (Zhizhu Kuanzhong Capsule) or the placebo group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Drug Group (Experimental): A 8-weeks double-blind treatment period with a Proprietary Chinese Medicine (consists of 4 kinds of Chinese herbs at 0.43g/capsule in weight), 3 capsules at one time, 3 times a day, oral administration 10-15 minutes before meals
  Interventions: Drug: Investigational drug for Functional Dyspepsia-Postprandial Distress Syndrome
- Placebo Group (Placebo Comparator): A 8-weeks double-blind treatment period with Placebo Capsules (at 0.43g/capsule in weight), 3 capsules at one time, 3 times a day, oral administration 10-15 minutes before meals
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Investigational drug for Functional Dyspepsia-Postprandial Distress Syndrome — The investigational drug is a new pure type of gastrointestinal function modulator traditional Chinese medicine, composed of 4 kinds of Chinese herbs: Rhizoma Atractylodis Macrocephalae, Fructus Aurantii Immaturus, Radix Bupleuri and Fructus Crataegi. The preliminary clinical trial showed that it has a good therapeutic effect on FD patients, its Fructus Aurantii Immaturus promotes gastric emptying by stimulating the cells to release motilin, thereby significantly improving patients' symptoms of fullness, epigastric pain, eructation, and nausea and vomiting.
  Other Names: Zhizhu Kuanzhong Capsule
  Arms: Investigational Drug Group
Drug: Placebo capsules — The placebo consist of mainly starch and microcrystalline cellulose, the usage and dosage are the same as the investigational drug.
  Other Names: Study drug
  Arms: Placebo Group

SUMMARY:
A 13 weeks randomized, double-blind and placebo parallel-controlled trial will be conducted to evaluate the clinical efficacy and safety of Zhizhu Kuanzhong Capsule in the treatment of functional dyspepsia-postprandial distress syndrome.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo parallel-controlled International clinical trial of Zhizhu Kuanzhong Capsule in treating patients with Functional Dyspepsia-Postprandial Distress Syndrome (FD-PDS).

In this study, Hong Kong Baptist University will collaborate with Xiyuan Hospital of China Academy of Chinese Medical Sciences, and will be recruiting 60 FD-PDS patients as study subjects in Hong Kong, out of the total sample size of 480 patients.

The study includes a 1 week run-in period, 8 weeks double-blind treatment period and a 4 weeks of follow up period for each eligible subject. Eligible subjects will be randomly assigned to either the trial drug or the placebo.

6 follow-up visits and 1 telephone follow-up will be scheduled for each subject on the -7 days (visit 1), enrollment on day 0 (visit 2), 14th day (visit 3), 28th day (visit 4), 42nd day (visit 5, telephone follow-up), the 56th day (visit 6) and the 84th day (visit 7) respectively.

Urine, stool and blood samples will be collected from each subject on visit 2 and visit 6 for blood, urine, stool, liver and kidney function tests.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the Rome IV diagnostic criteria for functional dyspepsia-postprandial distress syndrome;
2. At least 3 days during the one-week run-in period with VAS score ≥ 4 for major symptoms (at least one of postprandial fullness discomfort and early satiety) .
3. Be able to discontinue prohibited medications that may affect the evaluation of the effectiveness.
4. Written informed consent.

Exclusion Criteria:

1. Gastroscopic findings of gastric cancer, peptic ulcer, erosive gastritis (grade 2 or higher), moderate to severe atrophic gastritis, dysplasia, or other organ gastrointestinal disease.
2. History of abdominal surgery (except for appendectomy and cesarean section);
3. Immune system defects, or those who have been administered immunosuppressive agents or glucocorticoids within the past 3 months.
4. With combined severe cardiac and pulmonary insufficiency, insufficiency of liver (ALT/AST > 1.5 times the upper limit of the normal value), kidney insufficiency (BUN/SCr > the upper limit of the normal value), abnormal of endocrine system, abnormal hematopoietic system, and iron deficiency anemia as indicated on hematological examination.
5. With severe anxiety and depression.
6. With psychosis and mental retardation, language disorder precluding the ability of filling scales or recording symptoms.
7. Pregnancy or lactating; or patients of childbearing potential without effective contraception.
8. known to be allergic to the ingredients of this drug.
9. suspected or confirmed history of alcohol or drug abuse.
10. have participated in a clinical trial in the past 3 months.
11. deemed by the investigator as being not suitable for participation in the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) | For 8 weeks
  Subjects with the functional dyspepsia-postprandial distress syndrome are self-rated on the Visual Analogue Score (VAS) for the degree of discomfort with both symptoms of postprandial fullness and early fullness, with subjects indicating the degree of discomfort on a 10 cm ruler marked 0- "Asymptomatic or No Discomfort "and 10- "Extreme Severe or Extreme Discomfort "at its head and tail, respectively. The record is made on the diary card once a day and 7 days a week.
  The integral average for the sum of VAS for both two symptoms over the past week is evaluated based on the diary card content, and a 50% decrease from baseline in the integral average at 8 weeks is recorded as a response. The proportion of the response at 8 weeks after randomization is considered primary efficacy endpoint.

SECONDARY OUTCOMES:
Evaluation of individual symptoms of Functional Dyspepsia | For 8 weeks
  The subjects were evaluated using a symptom diary for Functional Dyspepsia based on the Visual Analogue Score (VAS) for gastrointestinal symptoms, including postprandial fullness discomfort, early satiety, abdominal distension, abdominal pain, epigastric burning sensation, nausea, excessive eructation, heartburn, vomiting, regurgitation, dysphagia, rass, abdominal enlargement, and defecation smoothness. Subjects indicated their discomfort on a 10 cm ruler marked 0-"asymptomatic or no discomfort" and 10-"very painful or extremely uncomfortable" on the head and tail respectively. The rating is made once a day and 7 days a week. The investigator used the average of the weekly VAS scores recorded in the subject's diary card as the symptom intensity score for this week, with one VAS score per week. The change of VAS score of each symptom at 8 weeks after randomization relative to the base
Overall Treatment Evaluation scale (OTE) | For 8 weeks
  The overall treatment efficacy is evaluated using a 7point Likert Overall Evaluation Scale (OTE). The clinical investigators asked the subjects the following questions at the visit: "In the last week, how much have your dyspeptic symptoms been alleviated as compared to pre-treatment?" There are 7 options: ① the symptoms improved significantly, ② the symptoms improved, ③ the symptoms improved slightly, ④ the symptoms did not change, ⑤ the symptoms aggravated slightly, ⑥ the symptoms aggravated, ⑦ the symptoms aggravated significantly. At the last visit time point of the treatment cycle, patients who selected ① -② were defined as treatment responders, and those who selected ③ -⑦ were defined as non-responders. The response rates at 8 weeks between the groups were compared for differences.
Hospital Anxiety and Depression Scale (HAD) score | At baseline, week 4 and week 8
  HAD Rating Scale scores are recorded at baseline, week 4 and week 8 during the double-blind treatment respectively. 14 questions are asked about the subject's emotional changes that best match his/her mood since the last month.
Short Form-Nepean Dyspepsia Index (SFNDI) | At baseline, week 4 and week 8
  Short Form-Nepean Dyspepsia Index (SFNDI) is recorded at baseline, week 4 and week 8 during the double-blind treatment respectively. 10 Questions are asked about how the subject's stomach pain, discomfort, or other epigastric symptoms over the last 14 days have affected his/her life.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxiang Bian, MD., Ph.D, Study Director — Hong Kong Chinese Medicine Clinical Study Centre
Locations (1):
- Linda Zhong, Kowloon Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided